CLINICAL TRIAL: NCT00068575
Title: A Phase II Trial of Pancreaticoduodenectomy Plus Postoperative Cisplatin, Interferon Alfa-2b, and 5-FU Combined With Radiation Treatment for Patients With Resected Pancreatic Adenocarcinoma
Brief Title: Chemotherapy, Interferon Alfa, and Radiation Therapy in Treating Patients Who Have Undergone Surgery For Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID02-040; P30CA016672 (NIH); MDA-ID-02040 (Other: UT MD Anderson Cancer Center); CDR0000327752 (Registry Identifier: NCI PDQ); NCT01053351 (obsolete NCT alias)
Record Dates: First submitted 2003-09-10; First posted 2003-09-11 (Estimated); Results first posted 2012-02-14 (Estimated); Last update posted 2012-02-15 (Estimated); Status verified 2012-02

CONDITIONS: Pancreatic Cancer
Keywords: stage I pancreatic cancer; stage II pancreatic cancer; stage III pancreatic cancer; adenocarcinoma of the pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Interferon-alpha; Interferon alpha-2; Cisplatin; Fluorouracil; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Postoperative Chemoradiation Regimen (Experimental): Postoperative Cisplatin 30 mg/m^2 intravenous (IV) weekly for 6 doses, Interferon Alfa-2b 3 million units subcutaneous (SQ) on Monday, Wednesday and Friday days 1-19 and 29-45 for 17 total doses, and 5-fluorouracil (5-FU) 175 mg/m2/day by continuous intravenous infusion days 1-19 and 29-45 with concurrent Radiation Treatment.
  Interventions: Biological: Recombinant Interferon Alfa; Drug: Cisplatin; Drug: Fluorouracil; Radiation: Radiation Therapy

INTERVENTIONS:
Biological: Recombinant Interferon Alfa — 3 million units subcutaneously every other day (Monday, Wednesday and Friday) during Days 1-19 and 29-45, for 6 1/2 weeks totaling 17 doses.
  Other Names: Interferon alfa-2b; IFN
Drug: Cisplatin — 30 mg/m^2 IV over 60 minutes on days 1, 8, 15, 29, 36, 43 - weekly for total 6 doses, during 5 1/2 weeks radiation therapy.
  Other Names: Platinol-AQ; Platinol; CDDP
Drug: Fluorouracil — 175 mg/m^2/day continuous infusion over 6 1/2 weeks for total 3 courses: Days 1-19 and 29-45, Days 71-108 and Days 127-168.
  Other Names: 5-fluorouracil; Adrucil; Efudex
Radiation: Radiation Therapy — External beam radiation on days 1-19 and days 29-45, 9 day treatment break on day 20.
  Other Names: RT; Radiatherapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cisplatin and fluorouracil, use different ways to stop tumor cells from dividing so they stop growing or die. Biological therapies such as interferon alfa may interfere with the growth of the tumor cells and slow the growth of cancer. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining chemotherapy and interferon alfa with radiation therapy after surgery may kill any remaining tumor cells.

PURPOSE: This phase II trial is studying how well giving cisplatin, fluorouracil, and interferon alfa together with radiation therapy works in treating patients who have undergone surgery for stage I, stage II, or stage III pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the overall survival of patients with previously resected pancreatic adenocarcinoma treated with postoperative cisplatin, interferon alfa, fluorouracil, and concurrent radiotherapy.
* Determine the toxic effects of this regimen in these patients.

Secondary

* Determine the disease-specific, biochemical failure-free, and symptom/treatment-free survival of patients treated with this regimen.
* Determine the quality of life of patients treated with this regimen.

OUTLINE:

* Chemoradiotherapy: Patients receive fluorouracil intravenous (IV) continuously and interferon alfa subcutaneously (SQ) 3 times per week (total of 17 doses) on days 1-19 and 29-45 and cisplatin IV over 6 hours on days 1, 8, 15, 29, 36 and 43. Patients also undergo concurrent radiotherapy once daily, 5 days a week in weeks 1-3 and 5-7 (28 fractions).
* Post-chemoradiotherapy fluorouracil: Patients receive fluorouracil IV continuously on days 71-108 and 127-168.

PROJECTED ACCRUAL: A total of 44 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy proven completely resected (R0 or R1) pancreatic adenocarcinoma of the pancreatic head or uncinate process [American Joint Committee on Cancer (AJCC) Stage I-III]. Surgery (pancreaticoduodenectomy) may be performed at M. D. Anderson Cancer Center or prior to referral to M. D. Anderson Cancer Center. Protocol treatment must begin within 12 weeks of surgery.
2. Postoperative (pre-treatment) computed tomography (CT) scan without evidence of radiographically defineable residual primary/metastatic disease or clinically significant post-surgical changes.
3. Staging studies completed within three weeks +/- 3 days of protocol registration.
4. Hemoglobin (Hb) >9.0 g/%, White Blood Count (WBC) >3,000 cells/mm3 (Absolute neutrophil count (ANC)>1,500 cells/mm3), platelets >75,000 cells/mm3.
5. Postoperative serum calcium (CA) 19-9 < 100.
6. Performance status: Zubrod 0 or 1.
7. Creatinine £1.5 mg/dL and calculated or measured creatinine clearance (CrCl) of 60 ml/min or greater by the following formula: Creatinine clearance rate (CrCl) = (140 - age) * Weight (kg) * 0.85 (female) OR * 1.00 (male) 72 * serum creatinine
8. Patients should have bilateral renal function, as determined on excretory urogram (IVP) or abdominal CT, or ³ 2/3 of one functioning kidney must be able to be shielded from the radiation beam.
9. No acute infections at the time of therapy initiation.
10. Women of childbearing potential must agree to practice adequate contraception and to refrain from breast feeding, as specified in the informed consent.
11. Patients must sign a study-specific consent form, which is attached to this protocol.
12. Patients with a prior history of non-pancreatic malignancy who are free of disease from their primary cancer may be eligible at the discretion of the study chair.

Exclusion Criteria:

1. Residual (clinical or CT definable) metastatic or incompletely resected local disease.
2. Patients with positive peritoneal cytology (for adenocarcinoma) detected at laparotomy for pancreaticoduodenectomy or as part of prior laparoscopic assessment of peritoneal cytology.
3. Patients with a history of hypersensitivity to interferon alfa-2b.
4. Patients with significant cardiovascular disease, such as unstable angina or congestive heart failure.
5. Pregnancy or breastfeeding.
6. Patients with severe pulmonary disease.
7. Children under the age of 18 are excluded (as the disease is rare and toxicity profile of this regimen untested in pediatric patients).
8. Presence or history of severe depression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2002-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter W. Pisters, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- M. D. Anderson Cancer Center at University of Texas, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: May 31, 2002 to January 14, 2010. All recruitment was done at UT MD Anderson Cancer Center.
Pre-assignment Details: Of the 29 participants who were enrolled, one patient dropped out prior to receiving study treatment.
Period: Overall Study
Arm/Group | Postoperative Chemoradiation Regimen
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Postoperative Chemoradiation Regimen
Number analyzed (Participants) | 28
Age Continuous [Median (Full Range); unit: years] | 60.5 [39 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Median Overall Survival (OS)
Description: Overall Survival defined overall survival time, measured from date of tissue diagnosis till disease progression or death.
Time Frame: Participants followed till disease progression or death (approximately 6 years)
Population: Analysis by protocol.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Postoperative Chemoradiation Regimen
Number analyzed (Participants) | 28
months | 42 [32.1 to 64.5]

ADVERSE EVENTS:
Time Frame: Toxicity assessed for participants while on 6 week chemoradiation treatment period with a one week break (equivalent 7 weeks). Data collected over 7 years and 4 months through on-going follow up.
Description: Only adverse events during treatment for Common Toxicity Criteria (CTC) Grade 3 events and above were collected. Toxicities graded by the National Cancer Institute (NCI) 1998 CTC.
Arm/Group | Postoperative Chemoradiation Regimen
Serious Adverse Events (participants affected / at risk) | 25/28
Other Adverse Events (participants affected / at risk) | 0/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Postoperative Chemoradiation Regimen (N=28)
Leukopenia (Blood and lymphatic system disorders) | 15
Lymphopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 12
Febrile (Non-neutropenic) (Infections and infestations) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Elevated alkaline phosphate (Metabolism and nutrition disorders) | 1
Elevated Alanine transaminase (ALT) (Metabolism and nutrition disorders) | 1
Abdominal Pain (Investigations) | 2
Fatigue (General disorders) | 8
Hand/foot syndrome (Skin and subcutaneous tissue disorders) | 1
Anorexia (Gastrointestinal disorders) | 8
Dehydration (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Nausea/Vomiting (Gastrointestinal disorders) | 2
Mucositis/Stomatitis (Gastrointestinal disorders) | 9
Abdominal abscess (General disorders) | 1
Overdose of interferon alfa-2b (IFN) (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No